CLINICAL TRIAL: NCT06986837
Title: Role of Inflammasome in Platelet Activation in Sickle Cell Disease Patient
Acronym: DrePlaquette
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RNI_2019/08; 2019-A03033-54 (Other: CHU de la Guadeloupe)
Record Dates: First submitted 2025-05-06; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: platelets; NLRP3; HMGB1; BTK
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — one blood collection will be realized during the annual follow up visit of the patients and during the screening visit for the controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients SS: Sixty SS patients
- Patients SC: Twenty SC patients
- Control group AA: Patients without hemoglobin disease

SUMMARY:
Sickle cell disease is characterized by chronic hemolytic anemia, painful crisis called vaso-occlusive crisis and chronic inflammation. Activated platelets of Sickle cell disease patients participated to both chronic inflammation and painful vaso-occlusive crisis .

The main aim of this study is to characterize the contribution of Nucleotide-binding domain Leucine Rich repeat containing Protein 3 inflammasome in platelets' activation in Sickle cell disease and to connect platelet activation, inflammation and sickle cell disease complication.

DETAILED DESCRIPTION:
During inflammation, platelets are activated through different cell signaling pathways, all of them leading to P selectin expression. Platelets activated by intravascular hemolysis (hemoglobin and heme) and High-Mobility Group Box protein 1 released by activated cells, participate to vaso-occlusive crisis occurrence through an increase of pro-inflammatory state. Toll-Like Receptor 4, expressed at the membrane of platelets, and the Nucleotide-binding domain Leucine Rich repeat containing Protein 3. inflammasome expressed by platelets, may also be involved in these processes. In addition, platelets express Bruton Tyrosine Kinase which could be activated through Nucleotide-binding domain Leucine Rich repeat containing Protein 3 and Toll-Like Receptor 4 pathways. These platelet cell signaling activation pathways related to inflammation, not well explored in Sickle cell disease, could connect platelet activation, inflammation and vaso-occlusive crisis . In this study, the collaborators will determine Nucleotide-binding domain Leucine Rich repeat containing Protein 3 activation state in platelets of Sickle cell disease patients.

Sickle cell disease patients will be recruited in the active file of the sickle cell center of Guadeloupe. Two groups of patients will be constituted: SS patients and SC patients. The control group will be patients who came for screening at the sickle cell center of Guadeloupe (University hospital of Guadeloupe, Pointe à Pitre).

Only one blood collection will be realized during the annual follow up visit of the patients and during the screening visit for the controls.

ELIGIBILITY:
Inclusion Criteria:

* patients with SS or SC Sickle cell disease
* diagnosis of SCD performed by electrophoresis or HPLC in a reference laboratory for hemoglobinopathies
* clinically in a steady state at inclusion (without complication in the last month and without transfusion in the three last months)
* patient followed up for Sickle cell disease at the sickle cell center of Guadeloupe (University hospital of Guadeloupe, Pointe à Pitre)
* patients who will provide written informed consent in accordance with the Declaration of Helsinki
* patients affiliated to national social security

Exclusion Criteria:

* - patients with hemoglobinopathy other than SS and SC Sickle cell disease
* patients with a transfusion therapy or on bleeding therapy for less than three months
* patients no affiliated to national social security
* pregnant or breastfeeding patients
* patients who will not provide written informed consent in accordance with the Declaration of Helsinki

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with sicke cell disease in a steady state at inclusion
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
platelets' Nucleotide-binding domain Leucine Rich repeat containing Protein 3 activation | Baseline
  flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: veronique Baccini, MD PhD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Chu de La Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koehl B, Claude L, Reminy K, Tarer V, Baccini V, Romana M, Colin-Aronovicz Y, Damaraju VL, Sawyer M, Peyrard T, Etienne-Julan M, Le Van Kim C, Azouzi S, Reininger L. Erythrocyte type 1 equilibrative nucleoside transporter expression in sickle cell disease and sickle cell trait. Br J Haematol. 2023 Mar;200(6):812-820. doi: 10.1111/bjh.18586. Epub 2022 Dec 4. PMID 36464247